CLINICAL TRIAL: NCT03737617
Title: Immunoglobulin Replacement Therapy for Immunoglobulin G Subclass 2 Deficient Patients With Bronchiectasis- A Proof of Concept Study
Brief Title: Immunoglobulin Replacement Therapy for Immunoglobulin G Subclass 2 Deficient Patients With Bronchiectasis
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Cant obtain IMP
Sponsor: University of Edinburgh (Other)
Collaborators: NHS Lothian (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IgG2CT001
Record Dates: First submitted 2017-07-19; First posted 2018-11-09 (Actual); Last update posted 2021-09-29 (Actual); Status verified 2021-09

CONDITIONS: Bronchiectasis; Immunoglobulin Subclass Deficiency
Keywords: Replacement therapy; Microbiology; Exacerbations; Bronchiectasis; Immunoglobulin G subclass 2
MeSH Terms: conditions — Bronchiectasis | interventions — Hizentra

STUDY DESIGN:
Intervention Model Description: 1 Group receiving active immunoglobulin replacement therapy
Masking Description: 1 group receiving standard care
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active arm (Experimental): Weekly subcutaneous immunoglobulin therapy (0.1g/Kg) Cuvitru 20% Injectable Solution for 1 Year
  Interventions: Drug: Cuvitru 20 % Injectable Solution
- Control (No Intervention): Standard Care arm without immunoglobulin replacement therapy

INTERVENTIONS:
Drug: Cuvitru 20 % Injectable Solution — Active
  Arms: Active arm

SUMMARY:
Bronchiectasis is a common chronic lung condition where patients have permanent airways damage leading to daily symptoms of cough, sputum production and recurrent respiratory tract infections.

Preliminary studies in our research group have found a severe deficiency of the immune system as a rare cause of bronchiectasis (called immunoglobulin G subclass 2 deficiency) and occurs in about 1 in 20 bronchiectasis patients. The pilot work shows that these patients have more chest infections and their lung function deteriorates more rapidly.

There are no trials to date to guide doctors to decide whether we should replace this deficiency from donated blood or not. The aim with treatment is to prevent disease progression and avoid the need for long term antibiotics.

This trial will help us understand how this treatment works and its acceptability to patients. This study will help us decide whether investigators should pursue future formalised trials in many centres throughout the UK and how investigators should evaluate such a treatment.

We are looking to recruit 20 patients to this study 10 of which will receive weekly replacement therapy and the remaining 10 will receive standard care.

DETAILED DESCRIPTION:
Background What is bronchiectasis? Bronchiectasis is a chronic disabling condition due to permanently inflamed and damaged airways with patients suffering chronic cough, chronic sputum production and recurrent infections affecting 4-6 per 1,000 populations in the UK.

Causes of bronchiectasis There are a variety of causes of bronchiectasis with past infection being the commonest cause (29-42%). In about 30-53% no cause can be identified in bronchiectasis. National guidelines recommend screening for causes that are potentially treatable including immune deficiency, allergic bronchopulmonary aspergillosis, active environmental bacterial infection and cystic fibrosis as they all have therapies that may alter the disease progression.

Immunoglobulins in bronchiectasis Immunoglobulin A (IgA) and Immunoglobulin G (IgG) are the most common antibodies found in the lung, where they opsonize pathogens and protect the body from infection together with neutrophils and macrophages. Most bronchiectasis patients show higher than normal IgG and IgA antibody levels, which reflects the high degree of recurrent lung infections and chronic inflammation.

IgG has four subclasses (1-4), which bind to and opsonize different kinds of antigens. IgG2 primarily binds polysaccharides and carbohydrates that are found in bacterial capsules, the cell wall in gram-positive bacteria and the O-antigen of lipopolysaccharides found on the outer membrane of gram-negative bacteria, which makes IgG2 an important part of bacterial clearance in the lung.

The frequency of IgG2 deficiency in the general healthy population lies between 2 to 20% (N = 106). Paediatric studies show IgG2 deficiency was the most frequent IgG subclass deficiency, and in their study 10% already had bronchiectasis.

Studies to date investigating the frequency of IgG2 deficiency in bronchiectasis have been small in 56, 65 and 89 patients with IgG2 subclass deficiency varying between 5 and 29%.

Hypothesis/Rationale Immunoglobulin replacement therapy is recommended for IgG deficiency such as common variable immunodeficiency or agammaglobulinaemia to reduce infections but there is international debate whether patients with IgG subclass deficiency should be offered such treatment.

The investigators hypothesis is that IgG replacement therapy will benefit IgG2 deficient patients with bronchiectasis by reducing the bacterial burden in the airways and reducing the time to first exacerbation and reducing the overall exacerbation frequency.

STUDY DESIGN This will be an open labelled proof of concept randomised controlled trial in 20 patients- 10 will receive weekly subcutaneous IgG replacement therapy for 52 weeks and the other group no added treatment to standard care.

The technician will be blinded to the patient's treatment. The investigators have chosen the minimum patients per group to assess study feasibility and endpoints on mechanism and efficacy will help on deciding the endpoint and power of this endpoint for a future Randomised Controlled Trial (RCT).

Patients will be assessed at the following time points.

BASELINE Following confirmation of eligibility, participants will be invited to attend a baseline visit (this must take place within 8 weeks of screening).

At the baseline visit, participants will be randomised to remain on standard care alone or to receive standard care plus 52 weekly infusions of Cuvitru.

A trial diary will be provided to participant of both groups and the following assessments will be made:

* 24 hour sputum sample
* Induced sputum sample
* Lung function assessment
* Incremental Shuttle Walk Test
* Blood samples (approximately 80 ml)
* Questionnaires
* Adverse Events
* Concomitant Medications
* Sample pot provided for 24 hour sputum sample (week 26)
* Pregnancy Test (women of child bearing potential only)

For those randomised to the interventional group, weight will be measured and training will be provided to permit self-administration of the IMP at home. The first infusion of IMP will take place at the baseline visit. Weekly infusion visits will continue to take place at the Royal Infirmary of Edinburgh until the participant has been deemed competent to self-administer at home. At such time, sufficient IMP (and contingency supply) will be dispensed to permit weekly infusions until the Week 13 visit.

WEEKLY All participants will complete their diary on at least a weekly basis to record adverse events, exacerbations and concomitant medications.

Once competent, participants randomised to IgG replacement therapy will self-administer a weekly infusion of IMP at home (7±2 days following previous infusion). The date of infusion will be recorded in the diary and the vial sticker attached to document IMP use.

WEEK 13 (IgG Replacement Therapy Group Only) Participants will be asked to attend the hospital for an infusion visit 13 weeks (±2 weeks) following the baseline visit. A pregnancy test will be repeated for women of childbearing potential. Self-administration competency will be assessed during IMP infusion. Used/partially used vials of IMP and needles will be returned to the research team for destruction according to local policy. A 3 month supply of IMP (with contingency, if required) and necessary consumables will be dispensed. The completed diary will be returned to the research team and a new diary issued.

WEEK 26

Participants will attend a visit at 26 weeks (±2 weeks) following baseline. The following assessment will take place:

* 24 hour sputum sample
* Induced sputum sample
* Lung function assessment
* Incremental Shuttle Walk Test (ISWT)
* Blood samples (approximately 80 ml)
* Questionnaires
* Adverse Events
* Concomitant Medications
* Sample pot provided for 24 sputum sample (week 52)

All participants will return their completed trial diary to the research team and be issued a new one.

For participants in the IgG replacement therapy group only, self-administration competency will be assessed during IMP infusion. A pregnancy test will be repeated for women of childbearing potential. Used/partially used vials of IMP and needles will be returned to the research team for destruction according to local policy. A 3 month supply of IMP (with contingency, if required) and necessary consumables will be dispensed.

WEEK 39 (IgG Replacement Therapy Group Only) Participants will be asked to attend the hospital for an infusion visit 39 weeks (±2 weeks) following the baseline visit. A pregnancy test will be repeated for women of childbearing potential. Self-administration competency will be assessed during IMP infusion. Used/partially used vials of IMP and needles will be returned to the research team for destruction according to local policy. A 3 month supply of IMP (with contingency, if required) and necessary consumables will be dispensed. The completed diary will be returned to the research team and a new diary issued.

WEEK 52

Participants will attend the final visit at 52 weeks (or at a maximum of 54 weeks) following baseline. The following assessment will take place:

* 24 hour sputum sample
* Induced sputum sample
* Lung function assessment
* Incremental Shuttle Walk Test (ISWT)
* Blood samples (approximately 80 ml)
* Questionnaires
* Adverse Events
* Concomitant Medications

All participants will return their completed trial diary to the research team.

For participants in the IgG replacement therapy group only, all trial equipment will be returned to the research team. All used/partially used vials of IMP and needles will be returned to the research team for destruction according to local policy.

FOLLOW-UP 4 weeks (to a maximum of 5 weeks) following the 52 week visit, the research team will contact the participant by telephone to record any adverse events that have taken place since the previous visit.

This telephone call will be the last contact from the research team. Participants will then return to routine clinical care.

ELIGIBILITY:
Inclusion criteria (need to meet all criteria below)

1. Bronchiectasis as the primary respiratory diagnosis.
2. Aged 18 years or older.
3. Bronchiectasis Severity Index >5 (0-4 mild; 5-8 moderate; >9 severe) or 3 or more exacerbations in the preceding year.
4. Patients with IgG2 deficiency<2.41g/L.
5. Able to provide written, informed consent
6. In the opinion of the research physician, the patient will be able to comply with the requirements of the trial protocol
7. Meets the co-enrolment criteria

Exclusion criteria (will be excluded if they have any item below)

1. Cystic fibrosis
2. Pregnancy or breast feeding
3. Women of childbearing potential not taking appropriate contraception. Acceptable contraception in women of childbearing age is a "highly effective" contraceptive measure as defined by the Clinical Trials Facilitation Group (http://www.hma.eu/fileadmin/dateien/Human_Medicines/01-About_HMA/Working_Groups/CTFG/2014_09_HMA_CTFG_Contraception.pdf) and includes combined (oestrogen and progesterone containing) or progesterone-only contraception associated with inhibition of ovulation, or intrauterine device or bilateral tubal occlusion. Contraception must be continued for a minimum of 30 days after the end of the IMP dosing schedule.
4. Active malignancy
5. Active co-morbid illness
6. Current smokers or ex-smokers less than 1 year
7. Known hypersensitivity to L-proline or Polysorbate 80
8. Known hyperprolinaemia type I or II
9. Known hypersensitivity to the IMP active substance or excipients (i.e. human normal immunoglobulin, Glyine or water for injections).
10. Severe IgA deficiency and a history of hypersensitivity to human immunoglobulin treatment
11. Known IgG1 deficiency
12. Known thrombophilic disorders or thrombotic events
13. Previously participated in this trial
14. Severe renal impairment (creatinine clearance of less than 30 ml/minute)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-08-05 (Estimated); Primary Completion 2024-08-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Change in sputum bacterial load | 52 weeks
  With IgG replacement therapy, does the sputum bacterial load change in treated versus untreated group
Proportion with bacterial load >=10(6) colony forming units/ml | 52 weeks
  With IgG replacement therapy, does the frequency with >=10(6) colony forming units/ml change in treated versus untreated group?

SECONDARY OUTCOMES:
Change in sputum colour | 26 and 52 weeks
  Does sputum colour change in treated versus untreated group?
Change in sputum volume | 26 and 52 weeks
  Does 24 hour sputum volume change in treated versus untreated group
Change in sputum microbiome diversity | 52 weeks
  Does Sputum microbiome change in treated versus untreated group
Change of forced expired volume in 1 second | 26 and 52 weeks
  Does forced expired volume in 1 second change in treated versus untreated group
Change of forced expired volume in 1 second % predicted | 26 and 52 weeks
  Does forced expired volume in 1 second change % predicted in treated versus untreated group
Change of forced vital capacity | 26 and 52 weeks
  Does forced vital capacity in treated versus untreated group
Change of forced vital capacity % predicted | 26 and 52 weeks
  Does forced vital capacity % predicted in treated versus untreated group
Change of incremental shuttle walk test | 26 and 52 weeks
  Does the incremental shuttle walk test change in treated versus untreated group
Change of cough related quality of life using Leicester Cough Questionnaire mean score | 26 and 52 weeks
  Does cough related quality of life change in treated versus untreated group using the Leicester Cough Questionnaire mean score (range 3-21)
Change of cough related quality of life using Leicester Cough Questionnaire with 1.3 Unit or greater improvement | 26 and 52 weeks
  Does cough related quality of life change in treated versus untreated group using the Leicester Cough Questionnaire proportion that have 1.3 or more Unit improvement (minimum clinically important difference)
Change of quality of life using St George's Respiratory Questionnaire with 4Unit or greater improvement | 26 and 52 weeks
  Does quality of life change in treated versus untreated group using the St George's Respiratory Questionnaire proportion that have 4 Unit or more improvement (minimum clinically important difference)
Change of quality of life using St George's Respiratory Questionnaire mean score | 26 and 52 weeks
  Does quality of life change in treated versus untreated group using the St George's Respiratory Questionnaire mean score (range 0-100)
Change of sputum myeloperoxidase | 26 and 52 weeks
  Does sputum myeloperoxidase change in treated versus untreated group
Change of sputum elastase | 26 and 52 weeks
  Does sputum elastase change in treated versus untreated group
Change of sputum interleukin 8 | 26 and 52 weeks
  Does sputum interleukin 8 change in treated versus untreated group
Change of total IgG and subclasses | 26 and 52 weeks
  Do serum IgG and subclasses change in treated versus untreated group
Change of serum white cell count | 26 and 52 weeks
  Do serum white cell count change in treated versus untreated group
Change of serum C reactive protein | 26 and 52 weeks
  Do serum C reactive protein change in treated versus untreated group
Change of serum erythrocyte sedimentation rate | 26 and 52 weeks
  Do serum erythrocyte sedimentation rate change in treated versus untreated group
Change of serum intercellular adhesion molecule 1 | 26 and 52 weeks
  Do serum intercellular adhesion molecule 1 change in treated versus untreated group
Change of phagocytosis and killing of Pseudomonas aeruginosa | 26 and 52 weeks
  Does peripheral blood neutrophil phagocytosis and killing of Pseudomonas aeruginosa change in treated versus untreated group
Change of phagocytosis and killing of Staphylococcus aureus | 26 and 52 weeks
  Does peripheral blood neutrophil phagocytosis and killing of Staphylococcus aureus change in treated versus untreated group
Proportion with specific antibody deficiency | Baseline
  Is there antibody deficiency with pneumococcal vaccination
Time to first exacerbation requiring antibiotic therapy | 52 weeks
  Is the time to first exacerbation requiring antibiotic therapy change in treated versus untreated group
Number of exacerbations | 52 weeks
  Does the number of exacerbations change in treated versus untreated group
Frequency of exacerbations | 52 weeks
  Does the mean exacerbations change in treated versus untreated group
Number of participants with side effects | 26 and 52 weeks
  What are the number of participants with side effects of IgG therapy
Compliance rates of IgG therapy | 26 and 52 weeks
  What are the compliance rates of IgG therapy
Completion rates of IgG therapy | 26 and 52 weeks
  What are the completion rates of IgG therapy

CONTACTS AND LOCATIONS:
Overall Officials: Adam T Hill, MBChB MD, Principal Investigator — NHS Lothian and University of Edinburgh
Locations (1):
- Royal Infirmary of Edinburgh, Edinburgh, United Kingdom

IPD SHARING:
Plan to Share IPD: No
No plan to share IPD- will present overall data